CLINICAL TRIAL: NCT02389153
Title: Feasability and Effectiveness of a Collaborative Care Intervention in the Secondary Prevention of Coronary Heart Disease - A Pilot Study
Brief Title: Feasability of Collaborative Care in the Secondary Prevention of Coronary Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Göttingen (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Principal Investigator, Christoph Herrmann-Lingen, Prof. Dr., University of Göttingen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Kollaborative Behandlung-01287; 01287 Kollaborative Behandlung (Other: IFS GmbH)
Record Dates: First submitted 2014-12-02; First posted 2015-03-17 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Coronary Heart Disease
Keywords: secondary prevention coronary heart disease; myocardial infarction; cardiovascular risk factors; collaborative care; quality of life; patients´ satisfaction with treatment
MeSH Terms: conditions — Coronary Disease; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- collaborative care, CHD (Experimental): Participants start with the collaborative care intervention at baseline directly after inclusion.
  Interventions: Behavioral: collaborative care CHD
- collaborative care CHD - waitlist (Active Comparator): Participants start with the intervention 6 months after baseline, in the meantime they receive tau.
  Interventions: Behavioral: collaborative care CHD

INTERVENTIONS:
Behavioral: collaborative care CHD — Over a time span of 6 months participants receive individualized treatment to reduce risk factors and improve quality of life, based on their preferences following a health plan, which they developed with their health coach.

SUMMARY:
The main focus of the pilot study is to evaluate the feasability and effectiveness of a collaborative care intervention for patients suffering from a coronary heart disease (CHD) with insufficient controlled health related risk factors in their lifestyle. The design of the study is a wait list control design. 30 patients will receive treatment immediately after submission, the other 30 after 6 months. An interdisciplinary team, including a care manager for each patient, will offer an individualized treatment plan, based on shared decision making for each patient to reduce risk factors and improve quality of life.

DETAILED DESCRIPTION:
The following assumptions will be evaluated:

1. The collaborative care concept is feasable in the context of the german health care system and leads to greater patient satisfaction
2. The team-based intervention leads to a decrease of cardiovascular risk factors of patients in the intervention group compared to participants in the waitlist condition
3. The collaborative care intervention leads to an improvement of quality of life as well as mental well being of participants in the intervention group compared to participants of the waitlist condition

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* coronary heart disease (angiographically oder clinically approved)
* sufficient knowledge of the german language
* at least one not sufficient controlled risk factor : Diabetes mellitus (HbA1c>7,5%), smoking, lack of physical activity (less than 60 minutes of light physical exercise per week), heightened stress level (PSS-4 >5), arterial hypertension (blood pressure despite medication repeatedly heightened >140/90 or in a 24-hour measurement >135/85 mmHg), hypercholesteremia (LDL >130 mg/dl)
* written informed consent to participate

Exclusion Criteria:

* no existence of an medically approved coronary heart disease
* insufficient knowledge of the german language and ulterior disabilities to complete the questionnaires or to understand the education about the Intervention
* existence of a psychosis
* drug dependency (except tobacco)
* dementia
* severe episode of Depression
* current suicidal tendency
* cardiac insufficiency NYHA 4
* missing informed consent
* malign tumor (unless curative treated and without relapse)
* acute coronary syndrome or cardiosurgery within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2017-11 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Patients´ satisfaction with treatment between baseline and the up to 12 months follow-up | up to 12 months follow-up
  September 2014: baseline for both groups; first 30 participants start with the Intervention, march 2015: 6-months follow-up for intervention group, participants from the wait list group start with active intervention phase, September 2015: 12-months follow-up intervention group; 6-months follow-up participants wait list group, march 2016: 12-months follow-up participants wait list group
Change in composite cardiovascular risk score | Baseline to six months
  Change in cardiovascular risk factor score comprised of secondary outcomes mentioned below

SECONDARY OUTCOMES:
Smoking | Baseline and up to 12 months follow-up
  Actual smoking behavior:yes
Lack of physical exercise | Baseline and up to 12 months follow-up
  Less than 60 minutes of light physical exercise per week
LDL cholesterol | Baseline and up to 12 months follow-up
  A LDL value of >130mg/dl or higher
Hypertension | Baseline and up to 12 months follow-up
  A blood pressure value of >140/90 mmHg or in a 24 hour measurement >135/85 mmHg
Increased HbA1c | Baseline and up to 12 months follow-up
  A HbA1c value of >7,5% or higher
Heightened level of stress | Baseline and up to 12 months follow-up
  A value in the PSS-4 >5 is an indicator for an heigtened stress level

OTHER OUTCOMES:
Physical strain | Baseline and up to 12 months follow-up
  Physical strain is measured with the 6-minutes walking test
Fear and depression | Baseline and up to 12 months follow-up
  Fear and Depression is measured with the HADS-D; Herrmann-Lingen, Buss & Snaith, 1995
Self-efficacy | Baseline and up to 12 months follow-up
  Self-efficacy is measured with the GSW-6; Romppel et al., 2006
Social support | Baseline and up to 12 months follow-up
  Social Support is measured with the ESSI-D, Cordes et al., 2009
Health-related quality of life | Baseline and up to 12 months follow-up
  Quality of life is measured with the SF-12, Radoschewski & Bellach,1999

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Herrmann-Lingen, Prof. Dr., Study Director — University of Goettingen, Department of Psychosomatic Medicine and Psychotherapy
Locations (1):
- Department of Psychosomatic Medicine and Psychotherapy, Univ. of Goettingen, Göttingen, Germany

REFERENCES:
- [Derived] Bosselmann L, Fangauf SV, Herbeck Belnap B, Chavanon ML, Nagel J, Neitzel C, Schertz A, Hummers E, Wachter R, Herrmann-Lingen C. Blended collaborative care in the secondary prevention of coronary heart disease improves risk factor control: Results of a randomised feasibility study. Eur J Cardiovasc Nurs. 2020 Feb;19(2):134-141. doi: 10.1177/1474515119880062. Epub 2019 Sep 28. PMID 31564125